CLINICAL TRIAL: NCT05026879
Title: Adverse Events Report of Inactivated COVID-19 Vaccine From 4040 Healthcare Workers
Brief Title: Adverse Events Report of Inactivated COVID-19 Vaccine
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Şeniz Akçay, Physical Medicine and Rehabilitation, Study Chair, Assoc. Prof., Bozyaka Training and Research Hospital
Other Study IDs: 24.02.2021-29
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; Vaccine Adverse Reaction
Keywords: COVID-19; Vaccine; Vaccination; Adverse effect
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Inactivated COVID-19 vaccine (CoronaVac) — The adverse events due to an inactivated COVID-19 vaccine.

SUMMARY:
Numerous vaccination studies are conducted to protect against COVID-19 infection, and preclinical and clinical studies are still ongoing worldwide. During this extraordinary period, the necessity to perform COVID-19 vaccine studies and immunization programs together has emerged. Many manufacturing companies have started mass production of vaccines accepting the risk of failure of vaccines during trials. Vaccine Adverse Effects (VAEs) need to be documented quickly. We aimed to determine the VAEs and to compare the frequency of VAEs between groups according to socio-demographic characteristics after the inactivated vaccine (Corona Vac®) was administered to healthcare workers (HCWs) in Turkey.

In this study, an online questionnaire was delivered to volunteer healthcare workers across the whole country. Sociodemographic characteristics, medical history, history of COVID-19 infection, and VAEs occurring after the first and second doses of inactivated vaccine were evaluated.

DETAILED DESCRIPTION:
A new coronavirus, severe acute respiratory syncytial coronavirus 2 (SARS-CoV-2) first appeared in China at the end of 2019 and attracted attention with clusters of pneumonia-like cases, which were later defined as coronavirus disease 2019 (COVID-19). Vaccine development is usually achieved over decades and therefore it is unprecedented to have access to such a large number of approved vaccines for COVID-19. In this process, great efforts were made by many organizations to cope with this pandemic that affected the whole world.

COVID-19 vaccines with different features in the form of vector-mediated, messenger RNA (mRNA) or inactivated vaccines are being produced worldwide. CoronaVac® is an inactivated vaccine against severe acute respiratory syncytial coronavirus 2 (SARS-CoV-2) developed by Sinovac Biotech, China which was approved by World Health Organization (WHO) in June 2021.

Vaccine Adverse Effect (VAE) is defined as "any adverse medical event that occurs after vaccination, which is thought to be due to a vaccine.

The primary endpoint of our study was to evaluate the VAEs reported after the first dose and the second doses following the inactivated vaccine (CoronaVac®), which was administered to HCWs in our country as a dose of 3 µg twice, 28 days apart. The secondary endpoint was the comparison of the frequency of VAE development between groups according to socio-demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

1)The HCWs vaccinated with two doses of CoronaVac.

Exclusion Criteria:

1. The HCWs under 18 years old
2. The HCWs those couldn't be able to complete the questionnaire accurately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The healthcare workers
Sampling Method: Non-Probability Sample
Enrollment: 4040 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-14 (Actual)

PRIMARY OUTCOMES:
Adverse events detection | 20 minutes
  An online questionnaire was delivered to obtain Vaccine Adverse Effects to volunteer Healthcare Workers in Turkey.

CONTACTS AND LOCATIONS:
Overall Officials: Selma Tosun, Prof., Principal Investigator — Izmir Bozyaka Education and Research Hospital; Hulya Ozkan Ozdemir, MD, Study Chair — Izmir Bozyaka Education and Research Hospital; Esin Erdogan, Assoc. Prof., Study Chair — University of Health Sciences, Izmir Bozyaka Education and Research Hospital; Seniz Akcay, Assoc. Prof., Study Chair — University of Health Sciences, Izmir Bozyaka Education and Research Hospital; Murat Aysin, Assis. Prof., Study Chair — Izmir Katip Celebi University, Faculty of Medicine; Neslihan Eskut, MD, Study Chair — University of Health Sciences, Izmir Bozyaka Education and Research Hospital; Pinar Ortan, Prof., Study Chair — University of Health Sciences, Izmir Bozyaka Education and Research Hospital; Burak Eskut, MD, Study Chair — University of Izmir Katip Celebi, Ataturk Education and Research Hospital
Locations (1):
- University of Health Sciences Izmir Bozyaka Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Huang DQ, Zou B, Yang H, Hui WZ, Rui F, Yee NTS, Liu C, Nerurkar SN, Kai JCY, Teng MLP, Li X, Zeng H, Borghi JA, Henry L, Cheung R, Nguyen MH. Epidemiology of COVID-19: A systematic review and meta-analysis of clinical characteristics, risk factors, and outcomes. J Med Virol. 2021 Mar;93(3):1449-1458. doi: 10.1002/jmv.26424. Epub 2020 Aug 25. PMID 32790106
- [Background] Gao Q, Bao L, Mao H, Wang L, Xu K, Yang M, Li Y, Zhu L, Wang N, Lv Z, Gao H, Ge X, Kan B, Hu Y, Liu J, Cai F, Jiang D, Yin Y, Qin C, Li J, Gong X, Lou X, Shi W, Wu D, Zhang H, Zhu L, Deng W, Li Y, Lu J, Li C, Wang X, Yin W, Zhang Y, Qin C. Development of an inactivated vaccine candidate for SARS-CoV-2. Science. 2020 Jul 3;369(6499):77-81. doi: 10.1126/science.abc1932. Epub 2020 May 6. PMID 32376603
- [Background] Xia S, Duan K, Zhang Y, Zhao D, Zhang H, Xie Z, Li X, Peng C, Zhang Y, Zhang W, Yang Y, Chen W, Gao X, You W, Wang X, Wang Z, Shi Z, Wang Y, Yang X, Zhang L, Huang L, Wang Q, Lu J, Yang Y, Guo J, Zhou W, Wan X, Wu C, Wang W, Huang S, Du J, Meng Z, Pan A, Yuan Z, Shen S, Guo W, Yang X. Effect of an Inactivated Vaccine Against SARS-CoV-2 on Safety and Immunogenicity Outcomes: Interim Analysis of 2 Randomized Clinical Trials. JAMA. 2020 Sep 8;324(10):951-960. doi: 10.1001/jama.2020.15543. PMID 32789505
- [Background] Che Y, Liu X, Pu Y, Zhou M, Zhao Z, Jiang R, Yin Z, Xu M, Yin Q, Wang J, Pu J, Zhao H, Zhang Y, Wang L, Jiang Y, Lei J, Zheng Y, Liao Y, Long R, Yu L, Cui P, Yang H, Zhang Y, Li J, Chen W, He Z, Ma K, Hong C, Li D, Jiang G, Liu D, Xu X, Fan S, Cheng C, Zhao H, Yang J, Li Y, Zou Y, Zhu Y, Zhou Y, Guo Y, Yang T, Chen H, Xie Z, Li C, Li Q. Randomized, Double-Blinded, Placebo-Controlled Phase 2 Trial of an Inactivated Severe Acute Respiratory Syndrome Coronavirus 2 Vaccine in Healthy Adults. Clin Infect Dis. 2021 Dec 6;73(11):e3949-e3955. doi: 10.1093/cid/ciaa1703. PMID 33165503
- [Background] Xia S, Zhang Y, Wang Y, Wang H, Yang Y, Gao GF, Tan W, Wu G, Xu M, Lou Z, Huang W, Xu W, Huang B, Wang H, Wang W, Zhang W, Li N, Xie Z, Ding L, You W, Zhao Y, Yang X, Liu Y, Wang Q, Huang L, Yang Y, Xu G, Luo B, Wang W, Liu P, Guo W, Yang X. Safety and immunogenicity of an inactivated SARS-CoV-2 vaccine, BBIBP-CorV: a randomised, double-blind, placebo-controlled, phase 1/2 trial. Lancet Infect Dis. 2021 Jan;21(1):39-51. doi: 10.1016/S1473-3099(20)30831-8. Epub 2020 Oct 15. PMID 33069281
- [Background] Zhang Y, Zeng G, Pan H, Li C, Hu Y, Chu K, Han W, Chen Z, Tang R, Yin W, Chen X, Hu Y, Liu X, Jiang C, Li J, Yang M, Song Y, Wang X, Gao Q, Zhu F. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine in healthy adults aged 18-59 years: a randomised, double-blind, placebo-controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Feb;21(2):181-192. doi: 10.1016/S1473-3099(20)30843-4. Epub 2020 Nov 17. PMID 33217362
- [Background] Wu Z, Hu Y, Xu M, Chen Z, Yang W, Jiang Z, Li M, Jin H, Cui G, Chen P, Wang L, Zhao G, Ding Y, Zhao Y, Yin W. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine (CoronaVac) in healthy adults aged 60 years and older: a randomised, double-blind, placebo-controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Jun;21(6):803-812. doi: 10.1016/S1473-3099(20)30987-7. Epub 2021 Feb 3. PMID 33548194